CLINICAL TRIAL: NCT00036647
Title: A Randomized Placebo Controlled Study of OSI-774 (Erlotinib HCl, Tarceva[TM]) in Patients With Incurable Stage IIIB/IV Non-small Cell Lung Cancer Who Have Failed Standard Therapy for Advanced or Metastatic Disease
Brief Title: OSI-774 (Tarceva) in Treating Patients With Stage III or Stage IV Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: OSI Pharmaceuticals (Industry)
Collaborators: Canadian Cancer Trials Group (Network)
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BR.21; NCT00026325 (obsolete NCT alias)
Record Dates: First submitted 2002-05-13; First posted 2002-05-14 (Estimated); Last update posted 2018-01-10 (Actual); Status verified 2015-06

CONDITIONS: Carcinoma, Non-small-cell Lung
Keywords: Non-Small Cell Lung Cancer; Tarceva; EGFR; erlotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Erlotinib Hydrochloride

INTERVENTIONS:
Drug: Tarceva (erlotinib HCl, OSI-774 )

SUMMARY:
The purpose of this study is to determine if OSI-774 will improve overall survival of patients with incurable stage IIIB/IV non-small cell lung cancer compared to standard of care. OSI-774 is a new type of drug under evaluation called an epidermal growth factor receptor (EGFR). OSI-774 is an investigational drug that has not yet been approved by the U.S. Food and Drug Administration (FDA).

ELIGIBILITY:
* Clinical diagnosis of stage IIIB or IV non-small cell lung cancer.
* Must have evidence of disease (clinical or radiological).
* Have failed 1 but no more than 2 prior chemotherapy regimens, have recovered from any side effects and have not had any chemotherapy for at least 21 days.
* If the patient has had surgery, the surgery was at least 2 weeks ago.
* Patients whose cancer has spread to their brain or central nervous system are eligible, providing that they have been on stable dose of steroids for at least 4 weeks and are free of symptoms.
* If the patient received radiation therapy, treatment was at least 4 weeks ago.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 731 (Actual)
Dates: Start 2001-11-01 (Actual); Primary Completion 2004-01-30 (Actual); Study Completion 2004-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frances Shephard, M.D., Principal Investigator — Princess Margaret Hospital, Canada
Locations (97):
- United States (2):
  - University of Chicago Medical Center, Chicago, Illinois
  - University of Washington, Seattle, Washington
- Argentina (7):
  - Centro Medico Confidence, Buenos Aires, CP
  - Hospital Britanico, Buenos Aires
  - Hospital Interzonal de Agudos Evita, Buenos Aires
  - Instituto Alexander fleming, Buenos Aires
  - Hospital Churruca Visca, Buenos Aires
  - Instituto Oncologico Angel Roffo, Capital Federal
  - Hospital Italiano, Capital Federal
- Australia (10):
  - Canberra Hospital- Australia, Woden, Australian Capital Territory
  - Prince of Wales Hospital, Randwick, New South Wales
  - Newcastle Mater Misericordiae Hospital, Waratah, New South Wales
  - Southern Medical Day Care Center, Wollongong, New South Wales
  - Western Hospital, Footscray, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
  - Royal Adelaide Hospital, South Australia
  - Peter MacCallum Cancer Institute, Victoria
  - Austin & Repatriation Medical Centre, Victoria
- Brazil (9):
  - Instituto do Cancer do Ceara, Fortaleza, CEP
  - Instituto Nacional de Cancerologia, Rio de Janeiro, CEP
  - Nucleo de Oncologia da Bahia, Salvador, Estado de Bahia
  - Hospital Vera Cruz S/A, Belo Horizonte, MG CEP
  - Irmandade Santa Casa de Miseicordia de Porto, Porto Alegre, RS CEP
  - Hospital Sao Lucas da PUCRS, Porto Alegre, RS CEP
  - Faculdade de Medicina do ABC, Santo André, SP CEP
  - Escola Paulista de Medicina, São Paulo, SP CEP
  - Instituto do Cancer Arnaldo Vieira de Carvalho, São Paulo, São Paulo
- Canada (27):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Cancer Centre for the Southern Interior, Kelowna, British Columbia
  - BCCA - Vancouver Island, Victoria, British Columbia
  - CancerCare Manitoba (CCMB), Winnipeg, Manitoba
  - Dr.H. Bliss Murphy Cancer Centre, St. John's, Newfoundland and Labrador
  - QEII Health Sciences Centre, Halifax, Nova Scotia
  - The Royal Victoria Hospital, Barrie, Ontario
  - Northeastern Ontario Regional Cancer Centre, Greater Sudbury, Ontario
  - Hamilton Regional Cancer Centre, Hamilton, Ontario
  - Kingston Regional Cancer Centre, Kingston, Ontario
  - Credit Valley Hospital, Missisauga, Ontario
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Ottawa Regional Cancer Centre, Ottawa, Ontario
  - Peterborough Regional Health Centre, Peterborough, Ontario
  - Hotel Dieu Health Sciences Hospital, Saint Catherines, Ontario
  - Group Health Centre, Sault Saint Marie, Ontario
  - Toronto East General Hospital, Toronto, Ontario
  - Toronto-Sunnybrook Reg.Canc.Center, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Humbar River Regional Hospital, Weston, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec
  - McGill University, Montreal, Quebec
  - Hopital Du Sacre - Coeur De Montreal, Montreal, Quebec
  - Hopital Laval, Ste-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
- Institution: Clinica Las Condes, Santiago, Chile
- China (2):
  - Pamela Youde Nethersole Easter Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
- Germany (5):
  - Lungenklinik Heckeshorn, Berlin
  - Asklepios Fachkiniken, Gauting
  - Zentrum fur pheulmologie und Thoraxchirurgie, Großhansdorf
  - Thoraxklinik Heidelberg, Heidelberg
  - Lungenklinik Hermer, Hermer
- Sotiria Hospital, Athens, Greece
- Israel (8):
  - Haemek Medical Center, Afula
  - RAMBAM Medical Center, Haifa
  - Rabin Medical Center Beilinson Campus, Petach-Tiqva
  - Rabin Medical Center Golda Campus, Petach-Tiqva
  - Kaplan Medical Center, Rehovot
  - Sourasky Medical Center Oncology Institute, Tel Aviv
  - Sheba Medical Center Oncology Day Care, Tel Litwinsky
  - Assaf Harofeh Medical Center, Ẕerifin
- Mexico (3):
  - Instituto Nacional de Cancerologia, Mexico City, CP
  - Centro Estatal de Cancerologia de Durango, Durango
  - Hospital Central Sur de Alta Especialidad, PEMEX, Mexico City
- New Zealand (2):
  - Wellington Hospital, Riddiford Street, Wellington Region
  - Greenlane Hospital - New Zealand, Auckland
- Romania (4):
  - Oncology Institute Bucharest, Bucharest
  - Oncology Institute Ion Chiricuta, Cluj-Napoca
  - Spitalul Universitar, Iași
  - Clinical County Hospital, Sibiu
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre - Singapore, Singapore
- South Africa (9):
  - Durban Oncology Centre, Westbridge, Durban
  - Die Wilgers Hospital, Lynnwood, Pretoria
  - Oncotherapy Dept, National Hospital, Bloemfontein
  - Sandton Oncology Centre, Parklands
  - Johannesburg Hospital, Parktown
  - Eastern Cape Oncology Centre, Port Elizabeth
  - Mary Potter Oncology Centre, Pretoria
  - University of Pretoria, Pretoria
  - Rosebank Clinic Oncology Unit, Rosebank
- Sweden (2):
  - Lund University Hospital, Lund
  - Sahlgrenska University Hospital, Lund
- Thailand (3):
  - Pramongkutklao Hospital, Phayathai, Bangkok
  - Div. of Med Onc. The National Cancer Institute of Thailand, Bangkok
  - Chiangmai University, Chiang Mai

REFERENCES:
- [Background] Shepherd FA, Rodrigues Pereira J, Ciuleanu T, Tan EH, Hirsh V, Thongprasert S, Campos D, Maoleekoonpiroj S, Smylie M, Martins R, van Kooten M, Dediu M, Findlay B, Tu D, Johnston D, Bezjak A, Clark G, Santabarbara P, Seymour L; National Cancer Institute of Canada Clinical Trials Group. Erlotinib in previously treated non-small-cell lung cancer. N Engl J Med. 2005 Jul 14;353(2):123-32. doi: 10.1056/NEJMoa050753. PMID 16014882
- [Background] Tsao MS, Sakurada A, Cutz JC, Zhu CQ, Kamel-Reid S, Squire J, Lorimer I, Zhang T, Liu N, Daneshmand M, Marrano P, da Cunha Santos G, Lagarde A, Richardson F, Seymour L, Whitehead M, Ding K, Pater J, Shepherd FA. Erlotinib in lung cancer - molecular and clinical predictors of outcome. N Engl J Med. 2005 Jul 14;353(2):133-44. doi: 10.1056/NEJMoa050736. PMID 16014883
- See also: Link to results on Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=63